CLINICAL TRIAL: NCT04306198
Title: Helical Blade vs Lag Screw Fixation for Cephalomedullary Nailing of Low Energy Intertrochanteric Hip Fractures: Are There Differences in the Failure Rate? A Prospective, Randomized Study
Brief Title: Helical Blade vs Lag Screw Fixation for Cephalomedullary Nailing of Low Energy Intertrochanteric Hip Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Traumatologico Dr. Teodoro Gebauer Weisser (Other)
Responsible Party: Principal Investigator, Tomas Amenabar MD, Tomas Amenabar Vial , Head of hip and pelvis department., Instituto Traumatologico Dr. Teodoro Gebauer Weisser
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1937
Record Dates: First submitted 2020-03-04; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Hip Fractures
Keywords: Hip fractures; Intertrochanteric fractures; Helical blade; Cut-out
MeSH Terms: conditions — Hip Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lag Screw (Active Comparator): Device: Trochanteric Fixation Nail (TFN) whit lag screw Surgical stabilization of intertrochanteric hip fractures using two different proximal fixation implants
  Interventions: Device: Osteosynthesis with Trochanteric Fixation Nail (TFN), using a lag screw as a proximal fixation.
- Helical Blade (Active Comparator): Device: Trochanteric Fixation Nail (TFN) whit helical blade Surgical stabilization of intertrochanteric hip fractures using two different proximal fixation implants
  Interventions: Device: Osteosynthesis with Trochanteric Fixation Nail (TFN), using a helical blade as a proximal fixation.

INTERVENTIONS:
Device: Osteosynthesis with Trochanteric Fixation Nail (TFN), using a lag screw as a proximal fixation. — Closed reduction and surgical stabilization of intertrochanteric hip fractures using Trochanteric Fixation Nail (TFN), with lag screw as proximal fixation
  Arms: Lag Screw
Device: Osteosynthesis with Trochanteric Fixation Nail (TFN), using a helical blade as a proximal fixation. — Closed reduction and surgical stabilization of intertrochanteric hip fractures using Trochanteric Fixation Nail (TFN), with helical blade as proximal fixation
  Arms: Helical Blade

SUMMARY:
The purpose of this study will be to compare the failure and complications rates of and orthopedic implant (Cephalomedullary Nail) fixed with two different options actually available: lag screw or helical blade.

The study population will be patient who have been diagnosed with an intertrochanteric hip fracture.

Hypothesis: Our hypothesis is that the helical blade will have a higher failure rate compared to the lag screw

DETAILED DESCRIPTION:
Hip fractures in the elderly are recognized worldwide as a major public health problem, its incidence is increasing and it is expected to have 6,26 million cases per year worldwide by 2050.

Surgical treatment is recognized as the best option in these patients because it allows early rehabilitation and decreases mortality and complications.

Currently, the fixation with a cephalomedullary nail is the most commonly used treatment, since it has some mechanical advantages compared to other fixation methods and achieves adequate stability allowing early weight bearing and rehabilitation with low failure rates.

Changes in the design of these implants have tried to reduce the failure rate. The main change has been the introduction of the helical blade for cephalic fixation, instead of a lag screw. The concept behind this modification is that the blade would have greater fixation to the bone and less risk of cut out, because it is supposed to compact the bone around the helical blade instead of removing it.

In spite of some biomechanical studies in cadaveric or artificial models validating this biomechanical advantage, clinical series have shown controversial results. Recently, retrospective clinical studies have shown similar results with the use of the helical blade, and even some studies have shown a higher failure rate compared to the sliding screw.

Currently there is no prospective evidence regarding the failure rate of these two fixation methods. Our objective is to contribute with solid evidence to solve this answer. That is why we have designed a prospective randomized study with strict inclusion criteria, follow up and radiographic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Low Energy Mechanism
* Hip fracture classified as 31.A1.2 - 31 A1.3 and 31.A2 in the AO classification (year 2018)

Exclusion Criteria:

* Medical contraindication to surgery
* A fracture due to malignancy
* Peri implant fractures
* Inability to walk before the fracture
* An inability to comply with rehabilitation
* Non-ambulatory pre-fracture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Implant Failure | 6 months
  Rate of cut out , cut through, varus collapse

SECONDARY OUTCOMES:
Complications | 3 weeks, 3 months , 6 months
  Rate of Infection and Non Union.
Parker Mobility score | 3 months , 6 months
  Score , Minimum value 0 , maximum value 9 , higher scores mean a better outcome.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cooper C, Campion G, Melton LJ 3rd. Hip fractures in the elderly: a world-wide projection. Osteoporos Int. 1992 Nov;2(6):285-9. doi: 10.1007/BF01623184. PMID 1421796
- [Result] Sommers MB, Roth C, Hall H, Kam BC, Ehmke LW, Krieg JC, Madey SM, Bottlang M. A laboratory model to evaluate cutout resistance of implants for pertrochanteric fracture fixation. J Orthop Trauma. 2004 Jul;18(6):361-8. doi: 10.1097/00005131-200407000-00006. PMID 15213501
- [Result] Al-Munajjed AA, Hammer J, Mayr E, Nerlich M, Lenich A. Biomechanical characterisation of osteosyntheses for proximal femur fractures: helical blade versus screw. Stud Health Technol Inform. 2008;133:1-10. PMID 18376008
- [Result] Ibrahim I, Appleton PT, Wixted JJ, DeAngelis JP, Rodriguez EK. Implant cut-out following cephalomedullary nailing of intertrochanteric femur fractures: Are helical blades to blame? Injury. 2019 Apr;50(4):926-930. doi: 10.1016/j.injury.2019.02.015. Epub 2019 Feb 20. PMID 30885393